CLINICAL TRIAL: NCT00251030
Title: A Study To Estimate The Effect Of Omeprazole On The Pharmacokinetics Of Nelfinavir In Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Jasper Clinic, Michigan (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4301024
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Nelfinavir; Omeprazole

INTERVENTIONS:
Drug: Nelfinavir and Omeprazole

SUMMARY:
To estimate the effects of omeprazole on the pharmacokinetics of nelfinavir in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 18 and 55 years.

Exclusion Criteria:

* Subjects with hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To estimate the effects of multiple doses of omeprazole on the steady-state pharmacokinetics of nelfinavir and M8 in healthy subjects

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the 625 mg formulation of nelfinavir when administered alone and with omeprazole

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kalamazoo, Michigan, United States